CLINICAL TRIAL: NCT02028832
Title: Pilot Study of Pediatric Integrative Medicine in Pediatric Oncology, General Pediatrics and Pediatric Cardiology
Brief Title: Pediatric Integrative Medicine Trial Pilot
Acronym: PIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Principal Investigator, Sunita Vohra, Professor, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PIM1
Record Dates: First submitted 2013-12-16; First posted 2014-01-07 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Pain; Nausea; Vomiting; Anxiety
Keywords: pain; nausea/vomiting; anxiety; complementary and alternative medicine; pediatric; oncology; cost-effectiveness
MeSH Terms: conditions — Pain; Nausea; Vomiting; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): Usual care provided to pediatric inpatients
  Interventions: Procedure: Usual care
- PIM consult and service provision (Experimental): Pediatric integrative medicine service (PIM) through which pediatric inpatients will have the option of supplementing their usual care with acupuncture/acupressure, massage, and/or reiki
  Interventions: Procedure: PIM consult and service provision; Procedure: Usual care

INTERVENTIONS:
Procedure: PIM consult and service provision — If service is requested, treatment options include acupuncture/acupressure, massage, and reiki
  Arms: PIM consult and service provision
Procedure: Usual care — Usual care consists of all conventional care options in pediatric oncology including medication and other therapies.

SUMMARY:
This study will investigate if adding complementary therapies such as acupuncture, massage and reiki to inpatient pediatric care is feasible and what the effects are on outcomes such as patient symptoms, cost, safety, satisfaction and length of stay.

DETAILED DESCRIPTION:
Study Objective: To determine if a pediatric integrative medicine (PIM) service is effective in reducing overall symptoms of pain, nausea/vomiting, and/or anxiety (PNVA), length of stay, and costs, in hospitalized children when compared to conventional care. In this context, "integrative" refers to a combined approach of complementary and conventional medical therapies in an evidence-based fashion.

Design: cluster trial; 2-arm controlled evaluation study in pediatric oncology, general pediatrics and pediatric cardiology. Intervention will be offered during a 6-month PIM period following a 6 month control period.

Population: Inclusion criteria: (i) In-patients in participating division and (ii) informed consent/assent. Exclusion criteria: (i) lack of parent participation, fluency in English, or informed consent

Intervention: Recommendations for specific CAM therapies will be determined by a staff PIM pediatrician. Any combination of the following CAM therapies (dose, duration, amount to be based on patient need as assessed by CAM provider, patient, and parent): acupuncture/acupressure, massage, Reiki; all are to be offered in addition to usual care.

Control: Usual care.

Outcomes: Primary outcome: feasibility (i.e enrollment); Secondary outcomes: (i) PNVA symptom management, (ii) need for conventional pharmacotherapy, (iii) adverse events; (iv) parent and health care provider satisfaction with care provided, v) length of stay; and vi) cost-effectiveness (analysis of this outcome to be limited to patients admitted for at least 2 days and for not more than 30 days).

Significance: To our knowledge, this study will be the first comparative effectiveness trial to assess the impact of PIM for hospitalized children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* (i) all children, aged 0-16 years, who are admitted to Pediatric Oncology, General Pediatrics and Pediatric Cardiology at the Stollery Children's Hospital, Edmonton, Canada who
* (ii) can communicate in English; and
* (iii) give informed consent/assent

Exclusion Criteria:

* (i) cannot communicate in English;
* (ii) lack of parent availability to participate; or
* iii) lack of informed consent.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 872 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Enrollment | up to 5 days
  Enrollment of study participants over length of study which will inform conduct of a larger study in this population

SECONDARY OUTCOMES:
Change in pain | up to 5 days
  For pre-verbal children: Faces, Legs, Activity, Cry, Consolability tool Verbal children: faces Pain Scale-Revised
Change in nausea/vomiting | up to 5 days
  Baxter Retching Faces scale
Change in anxiety | up to 5 days
  Pediatrics Anxiety Faces scale
Incidence of adverse events | up to 5 days
  BC Children's Hospital Patient Safety Questionnaire; Canadian Pediatric Trigger tool
Parent satisfaction with patient care | up to 5 days
  Hospital's standardized satisfaction survey; State-Trait Anxiety Invenvtory
Length of hospital stay | up to 5 days

OTHER OUTCOMES:
Resource Utilization/Cost | Analysis of this outcome to be limited to patients admitted for at least 2 days and for not more than 30 days
  Resource utilization and related costs will be compared between study arms

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- Stollery Childrens' Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided